CLINICAL TRIAL: NCT06309082
Title: Application of High-frequency Contrast-enhanced Ultrasound in Visual Evaluation of Microcirculation in Diabetic Foot Ulcers
Brief Title: Assessing Diabetic Foot Ulcer Microcirculation With High-frequency Contrast Enhanced Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: DFU
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic Foot Ulcers; High-Frequency Contrast-Enhanced Ultrasound; Microcirculation blood supply assessment; Amputation; Limb salvage
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Amputation, Surgical; Debridement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic foot ulcer limb salvage group: The patient was treated without amputation
  Interventions: Procedure: Debridement
- Diabetic foot ulcer without limb salvage group: The treatment option for the patient was amputation
  Interventions: Procedure: Amputation

INTERVENTIONS:
Procedure: Amputation — Amputation was performed on diabetic foot ulcer
  Groups: Diabetic foot ulcer without limb salvage group
Procedure: Debridement — Debridement of diabetic foot ulcers was performed
  Groups: Diabetic foot ulcer limb salvage group

SUMMARY:
The objective of this observational study is to investigate and validate the utility of high-frame-rate ultrasound imaging technology for dynamic observation of the blood perfusion process at the site of ulcer wounds in real-time, focusing on patients with Diabetic Foot Ulcers (DFU). The primary research questions it seeks to address are as follows:

* What are the dynamic characteristics of vascular dynamics at the site of ulcer wounds in patients with DFU under high-frame-rate ultrasound imaging?
* Is High-Frequency Contrast-Enhanced Ultrasound (H-CEUS) technology feasible for effectively visualizing the microcirculation of ulcer wounds in patients with DFU? Participants will Undergo high-frame-rate ultrasound imaging for real-time observation of blood perfusion dynamics at the site of ulcer wounds.

Researchers will compare ulcerated sites with normal sites to see whether the use of High-Frequency Contrast-Enhanced Ultrasound (H-CEUS) has any discernible impact on the visualization of microcirculation in ulcer wounds.

DETAILED DESCRIPTION:
1. Investigate H-CEUS abnormalities in microcirculation at DFU ulcer sites Conduct H-CEUS detection of blood vessels at ulcer sites for each participant. Qualitatively and quantitatively analyze differences in contrast enhancement time, intensity, uniformity, direction, and vessel morphology among different patient groups based on time-intensity curves. Compare H-CEUS indicators between DFU ulcer and normal sites, followed by single-factor and multi-factor logistic regression analysis to identify meaningful imaging indicators for diagnosing DFU and construct an H-CEUS score.
2. Correlate H-CEUS score with traditional measurement indicators Perform color Doppler ultrasound (CDU), laser Doppler perfusion monitoring (LDPM), and transcutaneous partial pressure of oxygen (TcPO2) measurements at ulcer sites for participants. Analyze the correlation between H-CEUS score and the aforementioned five traditional microcirculation assessment methods. This analysis aims to determine if H-CEUS effectively reflects the degree of ischemia in DFU patients' ulcerated limbs, providing a new, non-invasive assessment tool to assist physicians in accurately assessing ulcer severity and tissue damage, facilitating the formulation of individualized and effective treatment plans.
3. Construct and evaluate the limb salvage predictive model using H-CEUS Conduct a retrospective analysis of clinical data from hospitalized DFU patients, categorizing them into limb salvage and amputation groups. Compare baseline data, biochemical indicators, and data based on H-CEUS scores between the two groups. Utilize single-factor and multi-factor logistic regression analysis to identify amputation-related risk factors. Subsequently, employ a random forest algorithm to construct a model based on H-CEUS data to predict limb salvage in DFU patients. To further validate the accuracy and clinical utility of this predictive model, nomogram charts and decision curve analysis (DCA) will be created.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the diagnosis criteria for diabetes
2. They exhibit concurrent peripheral neuropathy and/or lower limb vascular lesions
3. The feet show varying degrees of infection, ulcers, and/or damage to deep tissues

Exclusion Criteria:

1. Other causes of inflammatory skin reactions (such as trauma, gout, acute neuropathic arthropathy, fibular fracture, thrombosis, venous congestion)
2. Exclusion of patients with impaired fasting glucose and abnormal glucose tolerance
3. Diabetes complicated by stasis dermatitis
4. Use of medications or substances affecting vascular conditions, such as vasoconstrictors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetes is the second most common chronic disease, following hypertension. Diabetic foot ulcers are a prevalent and severe complication among diabetic patients, resulting from peripheral neuropathy or vascular lesions caused by thickening of the arterial walls and narrowing of the lumen in the lower limbs. This condition can lead to foot infections, ulcers, or deep tissue damage. In the early stages of the disease, patients may not perceive any noticeable changes, experiencing occasional walking pain in the feet. Without proper attention, this can progress to ulcers, difficulty in walking, and even gangrene, causing necrosis of muscles and bone tissues. In severe cases, it may lead to amputation, posing a significant threat to the patient's health.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
H-CEUS score | baseline, pre-intervention
  Establishment of the H-CEUS Score: Single-factor and multi-factor logistic regression analyses will be performed on parameters obtained from H-CEUS. H-CEUS candidate parameters with statistically significant values (p < 0.05) will be selected. Finally, the diagnostic model's H-CEUS scoring formula will be built using the identified indicators. The H-CEUS score is calculated as follows: H-CEUS Score = val(Parameter1) * β1 + val(Parameter2) * β2 + ⋯ + val(Parameter n) * βn + Intercept Value. Here, "val" represents the CEUS parameter value, and "β" represents the regression coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital the First Affiliated Hospital, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No